CLINICAL TRIAL: NCT04869423
Title: Effects of Dog-assisted Therapy in Adolescents With Eating Disorders: a Controlled Trial.
Brief Title: Animal-Assisted Therapy in Adolescents With Eating Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Daniel Collado-Mateo (Other)
Collaborators: Purina España (Reg. Trademark of Nestle S.A.) (Unknown)
Responsible Party: Sponsor-Investigator, Daniel Collado-Mateo, Assistant Professor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAT_Eat_Disorders
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Eating Disorders in Adolescence; Eating Disorders; Anorexia Nervosa/Bulimia
Keywords: Dog-assisted intervention; Eating Disorder Symptom; Depression; Anxiety; Adolescent behavior and character; Health-related quality of life; Strength; Body composition; Treatment satisfaction
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia; Depression; Anxiety Disorders; Adolescent Behavior | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Two groups: one control and one experimental group
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in this group will simply continue with their daily living and therapies. Assessments will be conducted before and after the 7wk program but patients in this group will not take part in it
- Experimental group (Experimental): Participants in this group will take part in 7 dog-assisted therapy sessions (1 per week). This therapy will be added to their usual daily living and therapies. Assessments will be conducted before and after the 7-week program.
  Interventions: Behavioral: Dog-Assisted Therapy

INTERVENTIONS:
Behavioral: Dog-Assisted Therapy — During seven weeks patients will assist one time per week (1 hour). The therapy will be conducted by an expert psychologist. The intervention will consist of 7 weeks conducted once a week (50 minutes each session). It will include three parts: 1) a welcome part aimed to get in touch with the dog, 2) a main part, where participants will be taught basic notions about dog training and then try to train the dogs. In this part, the patients will perform different activities and exercises with the dog. 3) A closing part to say goodbye to the dogs.
  Other Names: animal-assisted therapy; animal-assisted intervention
  Arms: Experimental group

SUMMARY:
This study aims to improve eating disorders symptomatology, mental, psychosocial and physical health, quality of life, strength and body composition of adolescents with eating disorders by the development of a dog-assisted therapy program.

The current research will involve thirty-two patients distributed equally in a control and an experimental group. The intervention group will participate once a week in a dog-assisted therapy of seven weeks. Moreover, all the included patients will participate in an assessment session before and after the intervention to compare the effects of the dog-assisted therapy within and between groups in anxiety, depression, character, behavior, eating disorder evolution, health-related quality of life, treatment satisfaction, strength and body composition.

Based on previous studies on different populations, it is expected that, compared to the control group, the experimental group may experience a potential reduction in anxiety, depression and symptoms, while improving quality of life, strength, body composition and behavior.

DETAILED DESCRIPTION:
Animal-Assisted Therapies (AAT) have proved to increase self-esteem, social capacity and impulse control while reducing anxiety and depression. Thus, AAT could be an innovative and effective therapy to improve the mental, social and physical health of adolescents with eating disorders.

Based on previous studies on different populations, it is expected that, compared to the control group, the experimental group may experience a potential reduction in anxiety, depression and symptoms, while improving quality of life, strength, body composition and behavior.

Thirty-two adolescents, younger than 18 years and diagnosed with eating disorders from the University Hospital Niño Jesus will participate in this study. The informed consent must be signed to be included in the study.

The intervention will consist of 7 weeks conducted once a week (50 minutes each session). It will include three parts: 1) a welcome part aimed to get in touch with the dog, 2) a main part, where participants will be taught basic notions about dog training and then try to train the dogs. In this part, the patients will perform different activities and exercises with the dog. 3) A closing part to say goodbye to the dogs.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents in the Psychiatry and Psychology Service of the Niño Jesús University Hospital
* Patients diagnosed with eating disorders
* Adolescents with the willingness to participate and availability to assist
* Having read and signed the written informed consent.

Exclusion Criteria:

* Patients with dog-allergy or dog phobia
* Adolescents with a history of impulsive animal aggression

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Eating disorder symptoms | At baseline and inmediately after the intervention (within 7 days after the last session)
  Measured by the EDI-2 questionnaire to evaluate the evolution of anorexia nervosa and bulimia nervosa normal symptoms. The EDI 2 is a 91 item scale with 8 subscales - (Drive for thinness, Bulimia, body dissatisfaction, ineffectiveness, perfection, interpersonal distrust, interoceptive awareness and maturity fears.). Respondents rate each item from 5 (usually), to 0 (never). Higher scores mean more severe symptoms.
Changes in Health-related quality of life | At baseline and inmediately after the intervention (within 7 days after the last session)
  Measured by the Kidscreen-10, which consists of 10 items scored on a 5-point Likert scale. Scores range between 10 and 50, and a higher score means better health-related quality of life.

SECONDARY OUTCOMES:
Changes in Anxiety | At baseline and inmediately after the intervention (within 7 days after the last session)
  Measured by the STAI-C questionnaire. It includes two different scales, one to asses state anxiety (20 items) and the other one to evaluate trait anxiety (20 items) in Spanish adolescents. Each item is rated from 1 to 3 thus, scores in each sub-scales can range from a minimum of 20 to a maximum score of 60. Higher scores mean higher anxiety.
Changes in Depression | At baseline and inmediately after the intervention (within 7 days after the last session)
  Measured by the Children Depression Inventory with the included 27 items, each one with 3 options, from 0 (absence of symptoms) to 2 (severe symptoms). The total score ranges from 0-54. Higher scores mean higher depression.
Changes in Adolescent character | At baseline and inmediately after the intervention (within 7 days after the last session)
  Measured by the Temperament and Character Inventory-Revised. It consists of 240 items and 5 options for each one. It measures 4 temperaments, Novelty Seeking (NS), Harm Avoidance (HA), Reward Dependence (RD), and Persistence (PS), and three characters, Self-directedness (SD), Cooperativeness (CO), and Self-transcendence (ST). Each item is scored from 1 to 5 with higher scores meaning higher levels in each dimension.
Changes in Behavior | At baseline and inmediately after the intervention (within 7 days after the last session)
  Measured by the Child Behavior Checklist inside the Achenbach System of Empirically Based Assessment to assess adolescents' psychopathology. It consists of 113 items and the parents must complete it to evaluate emotional and behavioural problems in children and adolescents. It is scored from 0="not true" to 2="true". Raw scores range from 0 to 226. Higher scores mean a worse outcome.
Changes in Strength | At baseline and inmediately after the intervention (within 7 days after the last session)
  Measured by a handgrip dynamometer (Takei) to evaluate the maximum strength applied with the hand.
Changes in Body mass | At baseline and inmediately after the intervention (within 7 days after the last session)
  Assessed using a weighing device
Treatment satisfaction | Inmediately after the intervention (within 7 days after the last session)
  Measured by the treatment satisfaction scale (CRES-4) by Feixas i Viaplana et al., 2012, which consists of 3 dimensions. The score in each one ranges from 0 to 100 and the global score is the sum of the dimensions (from 0 to 300). Higher scores mean higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Collado-Mateo, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Niño Jesús University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nunez BM, Sanchez JF, Perez AML, Rincon LL, Garcia MF, Garcia IG, Berna MG, Mateo DC. Effects of Dog-assisted Therapy in Anxiety Symptoms of Female Adolescents With Eating Disorders: A Controlled Trial. Actas Esp Psiquiatr. 2025 Dec;53(6):1265-1273. doi: 10.62641/aep.v53i6.1919. PMID 41437761